CLINICAL TRIAL: NCT03976024
Title: Necrotizing Bacterial Dermohypodermitis-necrotizing Fasciitis (DHBN-FN) Mono- or Multi-microbial Streptococcus Beta-haemolytic: Study of Carriage in Patients and Their Entourage
Brief Title: Necrotizing Bacterial Dermohypodermitis-necrotizing Fasciitis Mono- or Multi-microbial Streptococcus Beta-haemolytic
Acronym: STREPTO-FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP180348
Record Dates: First submitted 2019-03-15; First posted 2019-06-05 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2019-12

CONDITIONS: Streptococcus Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHBN-FN arm (Experimental): Recruitment is planned in traditional hospitalization for DHBN-FN patients. Evaluation of streptococcal carriage by swab, pharyngeal, anal and perineal in patients hospitalized for a DHBN-FN at the end of hospitalization and 1 month after discharge from hospital during the reassessment consultation. Swabs made by the dermatologist.
  The carriage of streptococcus in patients living under the same roof as patients with DHBN-FN will be evaluated by pharyngeal swab, anal and perineal. If the family accepts, the carriage of streptococcus in persons living under the same roof as patients with DHBN-FN will be evaluated by pharyngeal, anal and perineal swab in consultation. These swabs will be made within 10 days of diagnosis of DHBN-FN of the index
  Interventions: Other: DHBN-FN arm
- Control arm (Erysipelas) (Active Comparator): Recruitment is planned in traditional hospitalization for patients with erysipelas.
  The carriage of streptococcus in patients with erysipelas will be evaluated by pharyngeal, anal and perineal swab on day 0 (admission).
  Interventions: Other: Control arm (Erysipelas)

INTERVENTIONS:
Other: DHBN-FN arm — DHBN-FN will be evaluated by pharyngeal swab, anal and perineal. If the family accepts, the carriage of streptococcus in persons living under the same roof as patients with DHBN-FN will be evaluated by pharyngeal, anal and perineal swab in consultation. These swabs will be made within 10 days of diagnosis of DHBN-FN of the index
  Arms: DHBN-FN arm
Other: Control arm (Erysipelas) — The carriage of streptococcus in patients with erysipelas will be evaluated by pharyngeal, anal and perineal swab on day 0 (admission).
  Arms: Control arm (Erysipelas)

SUMMARY:
The aim of the study is to evaluate streptococcal carriage by swab, pharyngeal, anal and perineal in patients with DHBN-FN, in the entourage living under the same roof as well as patients with erysipelas

The main hypothesis is the major role of chronic porting of patients and entourage in DHBN-FN to SBH.

Indeed, the chronic pharyngeal / anal / perineal carriage could be a gateway following a transient bacteremia for a DHBN-FN.

The transmission of germs from the surrounding to the patient plays a major role:

At the gateway level in the case of exogenous DHBN-FN At the origin of chronic carriage in the case of endogenous DHBN-FN Transmission of germs from the patient to the surrounding area also plays an important role in increasing the risk of invasive SBH infections in the surrounding area.

ELIGIBILITY:
Inclusion Criteria:

* Patient:
* Major patient hospitalized for a DHBN-FN or erysipelas (clinical diagnosis determined at the entrance).
* Signed informed consent.

Case contact

* person of major age living under the same roof as a patient who has had a DHBN-FN.
* Signed informed consent

Exclusion Criteria:

* Patient:
* Minor patient
* Immunosuppressed patient: active hematology, poorly controlled HIV, neutropenia (PNN <1000 / mm3).
* Patient under guardianship or curatorship
* Patient deprived of liberty by judicial or administrative decision
* Patient not affiliated to a social security scheme and not a beneficiary of such a scheme

Case contact

* Minor person
* Person under tutorship or curatorship
* Person deprived of liberty by judicial or administrative decision
* Person not affiliated with a social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of beta-hemolytic streptococcus in patients with DHBN-FN | Day 0
  Evaluation of streptococcal carriage by swab, pharyngeal, anal and perineal in patients hospitalized for a DHBN-FN . Swabs made by the dermatologist. The detection of beta-hemolytic streptococcus will be made by culture
Rate of beta-hemolytic streptococcus in patients with DHBN-FN | 1 month after hospitalization discharge
  Evaluation of streptococcal carriage by swab, pharyngeal, anal and perineal in patients hospitalized for a DHBN-FN . Swabs made by the dermatologist. The detection of beta-hemolytic streptococcus will be made by culture
Rate of beta-hemolytic streptococcus in patients with DHBN-FN | Day 30
  Evaluation of streptococcal carriage by swab, pharyngeal, anal and perineal in patients hospitalized for a DHBN-FN . Swabs made by the dermatologist. The detection of beta-hemolytic streptococcus will be made by culture

SECONDARY OUTCOMES:
Prevalence of SBH carriage at the time of diagnosis | Day 0, Day 10
Sites of SBH carriage at the time of diagnosis | Day 0, Day 10
Rate of beta-hemolytic streptococcus in patients with erysipelas | Day 0
  The carriage of streptococcus in patients with erysipelas will be evaluated by pharyngeal, anal and perineal swab on day 0.
Rate of beta-hemolytic streptococcus in patients living under the same roof as patients with DHBN-FN | Up to 10 Days
  The carriage of streptococcus in persons living under the same roof as patients with DHBN-FN will be evaluated by pharyngeal, anal and perineal swab in consultation. These swabs will be made within 10 days of diagnosis of DHBN-FN of the index.
Main factors of streptococcal virulence | Day 0, Day 10
  Analyze the main factors of streptococcal virulence by Streptococcal genome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHOSODOW, Professor, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Henri Mondor Hospital-AP-HP, Créteil, France

IPD SHARING:
Plan to Share IPD: No